CLINICAL TRIAL: NCT01087905
Title: Improving the Population-Wide Effectiveness of U.S. Tobacco Cessation Quitlines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Wisconsin Department of Health and Family Services (Other Government); Consumer Wellness Solutions (Industry); Department of Health and Human Services (U.S. Federal Agency); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: H2009-0074; 1RC1CA144382-01 (NIH)
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Results first posted 2013-04-24 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-10

CONDITIONS: Smoking; Smoking Cessation
Keywords: Smoking; Smoking cessation; Medication adherence
MeSH Terms: conditions — Smoking; Smoking Cessation; Medication Adherence | interventions — Tobacco Use Cessation Devices; Nicotine Chewing Gum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- 2 Weeks of Nicotine Patch Only, No CMAC (Active Comparator): Participants in this randomization arm received 2 weeks of nicotine patch and standard cessation counseling (but no Cognitive Medication Adherence Counseling)
  2 Weeks of Nicotine patch dosed as follows:
  If > 10 cigs/day: one 21 mg nicotine patch per day for 2 weeks
  If < or = 10 cigs/day: one 14 mg nicotine patch per day for 2 weeks
  Interventions: Drug: Nicotine patch
- 2 Weeks of Nicotine Patch Only plus CMAC (Active Comparator): Participants in this randomization arm received 2 weeks of nicotine patch and standard cessation counseling plus Cognitive Medication Adherence Counseling
  2 Weeks of Nicotine patch dosed as follows:
  If > 10 cigs/day: one 21 mg nicotine patch per day for 2 weeks
  If < or = 10 cigs/day: one 14 mg nicotine patch per day for 2 weeks
  Interventions: Drug: Nicotine patch; Behavioral: CMAC
- 2 Wks Nicotine Patch+Nic Gum, No CMAC (Active Comparator): Participants in this randomization arm received 2 weeks of nicotine patch plus nicotine gum and standard cessation counseling (but no Cognitive Medication Adherence Counseling)
  2 Weeks of Nicotine patch dosed as follows:
  If > 10 cigs/day: one 21 mg nicotine patch per day for 2 weeks
  If < or = 10 cigs/day: one 14 mg nicotine patch per day for 2 weeks
  2 Weeks of Nicotine gum dosed as follows:
  If < 25 cigs/day, 2 mg nicotine gum for 2 weeks, at least 5 pieces of oral NRT per day (maximum of 1 piece every 1-2 hours), unless this amount of use produces nicotine toxicity effects.
  If ≥ 25 cigs/day, 4 mg nicotine gum for 2 weeks, at least 5 pieces of oral NRT per day (maximum of 1 piece every 1-2 hours), unless this amount of use produces nicotine toxicity effects.
  Interventions: Drug: Nicotine patch; Drug: Nicotine gum
- 2 Wks Nicotine Patch+Nic Gum plus CMAC (Active Comparator): Participants in this randomization arm received 2 weeks of nicotine patch and nicotine gum plus standard cessation counseling and Cognitive Medication Adherence Counseling
  2 Weeks of Nicotine patch dosed as follows:
  If > 10 cigs/day: one 21 mg nicotine patch per day for 2 weeks
  If < or = 10 cigs/day: one 14 mg nicotine patch per day for 2 weeks
  2 Weeks of Nicotine gum dosed as follows:
  If < 25 cigs/day, 2 mg nicotine gum for 2 weeks, at least 5 pieces of oral NRT per day (maximum of 1 piece every 1-2 hours), unless this amount of use produces nicotine toxicity effects.
  If ≥ 25 cigs/day, 4 mg nicotine gum for 2 weeks, at least 5 pieces of oral NRT per day (maximum of 1 piece every 1-2 hours), unless this amount of use produces nicotine toxicity effects.
  Interventions: Drug: Nicotine patch; Drug: Nicotine gum; Behavioral: CMAC
- 6 Weeks of Nicotine Patch Only, No CMAC (Active Comparator): Participants in this randomization arm received 6 weeks of nicotine patch and standard cessation counseling (but no Cognitive Medication Adherence Counseling)
  6 Weeks of Nicotine patch dosed as follows:
  If > 10 cigs/day: one 21 mg nicotine patch per day for 6 weeks
  If < or = 10 cigs/day: one 14 mg nicotine patch per day for 6 weeks
  Interventions: Drug: Nicotine patch
- 6 Weeks of Nicotine Patch Only plus CMAC (Active Comparator): Participants in this randomization arm received 6 weeks of nicotine patch and standard cessation counseling plus Cognitive Medication Adherence Counseling
  6 Weeks of Nicotine patch dosed as follows:
  If > 10 cigs/day: one 21 mg nicotine patch per day for 6 weeks
  If < or = 10 cigs/day: one 14 mg nicotine patch per day for 6 weeks
  Interventions: Drug: Nicotine patch; Behavioral: CMAC
- 6 Wks Nicotine Patch+Nic Gum, No CMAC (Active Comparator): Participants in this randomization arm received 6 weeks of nicotine patch plus nicotine gum and standard cessation counseling (but no Cognitive Medication Adherence Counseling)
  6 Weeks of Nicotine patch dosed as follows:
  If > 10 cigs/day: one 21 mg nicotine patch per day for 6 weeks
  If < or = 10 cigs/day: one 14 mg nicotine patch per day for 6 weeks
  6 Weeks of Nicotine gum dosed as follows:
  If < 25 cigs/day, 2 mg nicotine gum for 6 weeks, at least 5 pieces of oral NRT per day (maximum of 1 piece every 1-2 hours), unless this amount of use produces nicotine toxicity effects.
  If ≥ 25 cigs/day, 4 mg nicotine gum for 6 weeks, at least 5 pieces of oral NRT per day (maximum of 1 piece every 1-2 hours), unless this amount of use produces nicotine toxicity effects.
  Interventions: Drug: Nicotine patch; Drug: Nicotine gum
- 6 Wks Nicotine Patch+Nic Gum plus CMAC (Active Comparator): Participants in this randomization arm received 6 weeks of nicotine patch and nicotine gum plus standard cessation counseling and Cognitive Medication Adherence Counseling
  6 Weeks of Nicotine patch dosed as follows:
  If > 10 cigs/day: one 21 mg nicotine patch per day for 6 weeks
  If < or = 10 cigs/day: one 14 mg nicotine patch per day for 6 weeks
  6 Weeks of Nicotine gum dosed as follows:
  If < 25 cigs/day, 2 mg nicotine gum for 6 weeks, at least 5 pieces of oral NRT per day (maximum of 1 piece every 1-2 hours), unless this amount of use produces nicotine toxicity effects.
  If ≥ 25 cigs/day, 4 mg nicotine gum for 6 weeks, at least 5 pieces of oral NRT per day (maximum of 1 piece every 1-2 hours), unless this amount of use produces nicotine toxicity effects.
  Interventions: Drug: Nicotine patch; Drug: Nicotine gum; Behavioral: CMAC

INTERVENTIONS:
Drug: Nicotine patch — If > 10 cigs/day: one 21 mg nicotine patch per day
  If < or = 10 cigs/day: one 14 mg nicotine patch per day
Drug: Nicotine gum — If < 25 cigs/day, 2 mg nicotine gum, at least 5 pieces of oral NRT per day (maximum of 1 piece every 1-2 hours), unless this amount of use produces nicotine toxicity effects.
  If ≥ 25 cigs/day, 4 mg nicotine gum, at least 5 pieces of oral NRT per day (maximum of 1 piece every 1-2 hours), unless this amount of use produces nicotine toxicity effects.
  Other Names: Nicotine polacrilex
  Arms: 2 Wks Nicotine Patch+Nic Gum plus CMAC; 2 Wks Nicotine Patch+Nic Gum, No CMAC; 6 Wks Nicotine Patch+Nic Gum plus CMAC; 6 Wks Nicotine Patch+Nic Gum, No CMAC
Behavioral: CMAC — CMAC consists of tailored cessation counseling to improve medication adherence during the counseling calls. The CMAC protocol was developed by study investigators and involved: (1) pre-quit assessment of beliefs that might undermine NRT adherence; (2) on-going medication adherence assessment by quitline Quit Coaches; and (3) tailored coaching based on the ongoing assessments.
  Other Names: Cognitive Medication Adherence Counseling
  Arms: 2 Weeks of Nicotine Patch Only plus CMAC; 2 Wks Nicotine Patch+Nic Gum plus CMAC; 6 Weeks of Nicotine Patch Only plus CMAC; 6 Wks Nicotine Patch+Nic Gum plus CMAC

SUMMARY:
Research shows that smoking cessation is the most significant preventable health behavior change that a person can make to lower cancer risk. In addition, telephone quitlines are an effective, science-based smoking cessation treatment that is universally accessible to smokers in the U.S. However, little research has explored promising approaches that could increase quitline use, improve quit rates, and inform resource allocation for quitline services. The proposed study will test three promising enhancements to the standard quitline treatment that typically consists of counseling and, possibly 2 weeks of a NRT medication. These enhancements are: 1) combination nicotine replacement therapy as recommended by the United States Public Health Service Clinical Practice Guideline on Treating Tobacco Use and Dependence; 2) extended duration of cessation medication use; and 3) an innovative counseling addition - cognitive medication adherence counseling - to optimize adherence to cessation medication. In addition, the cost-effectiveness of each intervention will be calculated. The findings of the proposed research have broad potential application and relevance to state quitlines, quitline service providers, and other purchasers of quitline services such as employers and insurers. Additionally, the study findings can potentially inform other telephone health behavior counseling programs.

DETAILED DESCRIPTION:
The study design is a fully crossed 2x2x2 factorial design that tested the effect of two versus six weeks of nicotine replacement therapy (NRT), the effect of NRT monotherapy (nicotine patch alone) versus NRT combination therapy (nicotine patch + oral NRT), and the effect of cognitive medication adherence counseling (CMAC) versus no CMAC. A total of 987 smokers seeking cessation assistance from the Wisconsin Tobacco Quit Line (WTQL) were randomly assigned to the eight (2x2x2) different conditions generated by the three experimental factors. This design provides us with sufficient power to analyze each of our three main effects listed above. We will also test for two- and three-way interactions, but do not have sufficient data to make a priori assumptions about interaction effects. Finally, we will conduct a cost-effectiveness analysis for each of the three interventions to allow readers of this research to evaluate whether the additional costs of the interventions yield sufficient gains to warrant implementing them broadly.

ELIGIBILITY:
The only people eligible for this study are Wisconsin residents who contact the Wisconsin Tobacco Quit Line for smoking cessation services.

Inclusion Criteria:

* Callers will be eligible to participate in the study if they are English speaking; are 18 years of age or older; smoke a minimum of 10 cigarettes per day; are interested in quitting and are willing to set a quit date; willing and able to use nicotine patch and nicotine gum; agree to receive four follow-up counseling calls from Free & Clear (the quitline vendor for the State of Wisconsin); provide verbal informed consent; and provide contact information and agree to take four study follow-up calls from staff at the University of Wisconsin Center for Tobacco Research and Intervention.

Exclusion Criteria:

* Callers will be excluded if they are under the age of 18; are pregnant or breastfeeding; exclusively use other forms of tobacco (e.g., smokeless tobacco); are unwilling or unable to use study NRT medications; are currently using a cessation medication (NRT, bupropion, varenicline); or have medical exclusions as per FDA-approved product labeling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 987 (Actual)
Dates: Start 2010-04; Primary Completion 2011-02 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stevens S Smith, PhD, Principal Investigator — University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health; Paula A Keller, MPH, Study Director — University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health
Locations (2):
- United States (2):
  - Wisconsin Tobacco Quit Line (service provided by Free & Clear, Inc.), Seattle, Washington
  - University of Wisconsin Center for Tobacco Research and Intervention, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Upon request, clinical trial data will be shared with other investigators in the form of de-identified datasets. Requests can be sent to Stevens S. Smith, Ph.D., at sss@ctri.wisc.edu

REFERENCES:
- [Result] Smith SS, Keller PA, Kobinsky KH, Baker TB, Fraser DL, Bush T, Magnusson B, Zbikowski SM, McAfee TA, Fiore MC. Enhancing tobacco quitline effectiveness: identifying a superior pharmacotherapy adjuvant. Nicotine Tob Res. 2013 Mar;15(3):718-28. doi: 10.1093/ntr/nts186. Epub 2012 Sep 19. PMID 22992296
- See also: University of Wisconsin Center for Tobacco Research and Intervention — http://www.ctri.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult smokers who called the Wisconsin Tobacco Quit Line (WTQL) from April 1, 2010 to June 15, 2010 were invited to participate in the study; no advertising or targeted recruitment was utilized.
Groups:
- 2 Weeks of Nicotine Patch Only, No CMAC: Participants in this randomization group received 2 weeks of nicotine patch only and standard quitline cessation counseling consisting of 4 proactive counseling calls (but no Cognitive Medication Adherence Counseling (CMAC).
- 2 Weeks of Nicotine Patch Only Plus CMAC: Participants in this randomization group received 2 weeks of nicotine patch only and standard quitline cessation counseling consisting of 4 proactive counseling calls plus Cognitive Medication Adherence Counseling (CMAC).
- 2 Weeks of Nicotine Patch+Nicotine Gum , No CMAC: Participants in this randomization group received 2 weeks of nicotine patch plus nicotine gum and standard quitline cessation counseling consisting of 4 proactive counseling calls (but no Cognitive Medication Adherence Counseling (CMAC).
- 2 Weeks of Nicotine Patch+Nicotine Gum and CMAC: Participants in this randomization group received 2 weeks of nicotine patch plus nicotine gum and standard quitline cessation counseling consisting of 4 proactive counseling calls plus Cognitive Medication Adherence Counseling (CMAC).
- 6 Weeks of Nicotine Patch Only, No CMAC: Participants in this randomization group received 6 weeks of nicotine patch only and standard quitline cessation counseling consisting of 4 proactive counseling calls (but no Cognitive Medication Adherence Counseling (CMAC).
- 6 Weeks of Nicotine Patch Only Plus CMAC: Participants in this randomization group received 6 weeks of nicotine patch only and standard quitline cessation counseling consisting of 4 proactive counseling calls plus Cognitive Medication Adherence Counseling (CMAC).
- 6 Weeks of Nicotine Patch+Nicotine Gum , No CMAC: Participants in this randomization group received 6 weeks of nicotine patch plus nicotine gum and standard quitline cessation counseling consisting of 4 proactive counseling calls (but no Cognitive Medication Adherence Counseling (CMAC).
- 6 Weeks of Nicotine Patch+Nicotine Gum and CMAC: Participants in this randomization group received 6 weeks of nicotine patch plus nicotine gum and standard quitline cessation counseling consisting of 4 proactive counseling calls plus Cognitive Medication Adherence Counseling (CMAC).
Period: Overall Study
Arm/Group | 2 Weeks of Nicotine Patch Only, No CMAC | 2 Weeks of Nicotine Patch Only Plus CMAC | 2 Weeks of Nicotine Patch+Nicotine Gum , No CMAC | 2 Weeks of Nicotine Patch+Nicotine Gum and CMAC | 6 Weeks of Nicotine Patch Only, No CMAC | 6 Weeks of Nicotine Patch Only Plus CMAC | 6 Weeks of Nicotine Patch+Nicotine Gum , No CMAC | 6 Weeks of Nicotine Patch+Nicotine Gum and CMAC
Started | 119 | 126 | 123 | 122 | 122 | 127 | 121 | 127
Completed | 90 | 94 | 101 | 86 | 91 | 99 | 98 | 98
Not Completed | 29 | 32 | 22 | 36 | 31 | 28 | 23 | 29
Not completed — Lost to Follow-up | 24 | 28 | 18 | 31 | 27 | 25 | 20 | 24
Not completed — Withdrawal by Subject | 5 | 4 | 4 | 5 | 4 | 3 | 3 | 5

BASELINE CHARACTERISTICS:
Population: Baseline sample=987 adult smokers (at least 18 years of age) who called the Wisconsin Tobacco Quit Line (WTQL) from April 1, 2010 to June 15, 2010.
Groups:
- Total: Total of all reporting groups
Arm/Group | 2 Weeks of Nicotine Patch Only, No CMAC | 2 Weeks of Nicotine Patch Only Plus CMAC | 2 Weeks of Nicotine Patch+Nicotine Gum , No CMAC | 2 Weeks of Nicotine Patch+Nicotine Gum and CMAC | 6 Weeks of Nicotine Patch Only, No CMAC | 6 Weeks of Nicotine Patch Only Plus CMAC | 6 Weeks of Nicotine Patch+Nicotine Gum , No CMAC | 6 Weeks of Nicotine Patch+Nicotine Gum and CMAC | Total
Number analyzed (Participants) | 119 | 126 | 123 | 122 | 122 | 127 | 121 | 127 | 987
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
  Between 18 and 65 years | 115 | 119 | 121 | 119 | 116 | 119 | 114 | 123 | 946
  >=65 years | 4 | 7 | 2 | 2 | 6 | 8 | 6 | 4 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.33 (12.99) | 43.35 (12.61) | 41.39 (11.24) | 40.84 (11.96) | 41.74 (14.19) | 43.18 (13.627) | 42.61 (13.51) | 40.03 (13.31) | 41.93 (12.96)
Gender [Count of Participants; unit: Participants]
  Female | 71 | 65 | 63 | 70 | 75 | 72 | 74 | 79 | 569
  Male | 48 | 61 | 60 | 52 | 47 | 55 | 47 | 48 | 418
Region of Enrollment [Number; unit: participants]
  United States | 119 | 126 | 123 | 122 | 122 | 127 | 121 | 127 | 987

OUTCOME MEASURES:

1. Primary Outcome: 7-Day Point Prevalence Abstinence From Smoking by Intervention
Description: Self-reported total abstinence from any tobacco use (even a single puff) for the seven days preceding the target follow-up day.
Time Frame: 26 weeks after the target quit smoking date
Population: The study was originally powered to detect at least a 6.4% increase in the abstinence rate due to an enhanced intervention (e.g., 6 wks NRT); this effect size was based on prior quitline studies; we predicted that abstinence rates at 6 months would be approximately 12% in a standard intervention vs. 18.4% in an enhanced intervention.
Measure: Number; unit: Percentage of participants not smoking
Groups:
- Two Weeks of Nicotine Replacement Therapy (NRT): Participants in this intervention group received a two-week supply of Nicotine Replacement Therapy (NRT). This intervention is considered to be the standard intervention in terms of duration of NRT; it will be compared to the enhanced NRT duration intervention which is six weeks of NRT. Approximately half the total sample was randomized to the standard intervention (two weeks of NRT) and half to the enhanced intervention (six weeks of NRT).
- Six Weeks of Nicotine Replacement Therapy (NRT): Participants in this intervention group received a six-week supply of Nicotine Replacement Therapy (NRT). This intervention is considered to be the enhanced intervention in terms of duration of NRT; it will be compared to the standard NRT duration intervention which is two weeks of NRT. Approximately half the total sample was randomized to the standard intervention (two weeks of NRT) and half to the enhanced intervention (six weeks of NRT).
- NRT Monotherapy (Nicotine Patch Only): Participants in this intervention group received a single Nicotine Replacement Therapy (NRT) consisting of the Nicotine Patch only. This intervention is considered to be the standard intervention in terms of type of NRT; it will be compared to the enhanced NRT type intervention which is combination NRT consisting of Nicotine Patch plus Nicotine Gum (Combo NRT). Approximately half the total sample was randomized to the standard intervention (Nicotine Patch Only) and half to the enhanced intervention (Nicotine Patch plus Nicotine Gum).
- NRT Combination Therapy (Nicotine Patch Plus Nicotine Gum): Participants in this intervention group received Combination Nicotine Replacement Therapy (NRT) consisting of the Nicotine Patch plus Nicotine Gum. This intervention is considered to be the enhanced intervention in terms of type of NRT; it will be compared to the standard NRT type intervention which is NRT Monotherapy consisting of the Nicotine Patch Only. Approximately half the total sample was randomized to the standard intervention (Nicotine Patch Only) and half to the enhanced intervention (Nicotine Patch plus Nicotine Gum).
- Standard Cessation Counseling (No CMAC): Participants in this intervention group received standard quitline cessation counseling consisting of 4 proactive counseling calls. This intervention is considered to be the standard intervention in terms of cessation counseling; it will be compared to the enhanced cessation counseling intervention which consists of Standard Cessation Counseling plus Cognitive Medication Adherence Counseling (CMAC). Approximately half the total sample was randomized to the standard intervention (Standard Cessation Counseling, No CMAC) and half to the enhanced intervention (Standard Cessation Counseling plus CMAC).
- Standard Cessation Counseling Plus CMAC): Participants in this intervention group received standard quitline cessation counseling consisting of 4 proactive counseling calls plus Cognitive Medication Adherence Counseling (CMAC). This intervention is considered to be the enhanced intervention in terms of cessation counseling; it will be compared to the standard cessation counseling intervention which consists of Standard Cessation Counseling only (no CMAC). Approximately half the total sample was randomized to the standard intervention (Standard Cessation Counseling, No CMAC) and half to the enhanced intervention (Standard Cessation Counseling plus CMAC).
Arm/Group | Two Weeks of Nicotine Replacement Therapy (NRT) | Six Weeks of Nicotine Replacement Therapy (NRT) | NRT Monotherapy (Nicotine Patch Only) | NRT Combination Therapy (Nicotine Patch Plus Nicotine Gum) | Standard Cessation Counseling (No CMAC) | Standard Cessation Counseling Plus CMAC)
Number analyzed (Participants) | 490 | 497 | 494 | 493 | 485 | 502
Percentage of participants not smoking | 43.3 | 48.9 | 42.3 | 49.9 | 47.6 | 44.6
Statistical Analysis 1: Comparison: Two Weeks of Nicotine Replacement Therapy (NRT) vs NRT Monotherapy (Nicotine Patch Only); Null hypothesis: No difference in abstinence rates for participants receiving Two Weeks of Nicotine Replacement Therapy (NRT) versus Six Weeks of Nicotine Replacement Therapy (NRT). We hypothesized that Six Weeks of NRT would result in statistically significantly higher abstinence rates compared to Two Weeks of NRT. The study was originally powered to detect at least a 6.4% increase in the abstinence rate due to an enhanced intervention (e.g., 6 wks NRT); Test type: Superiority or Other; p = .076, Regression, Logistic; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.98 to 1.61]
Statistical Analysis 2: Comparison: NRT Monotherapy (Nicotine Patch Only) vs NRT Combination Therapy (Nicotine Patch Plus Nicotine Gum); Null hypothesis: No difference in abstinence rates for participants receiving NRT Monotherapy (Nicotine Patch Only) versus NRT Combination Therapy (Nicotine Patch plus Nicotine Gum). We hypothesized that Combination NRT would result in statistically significantly higher abstinence rates compared to NRT Monotherapy. The study was originally powered to detect at least a 6.4% increase in the abstinence rate due to an enhanced intervention (e.g., Combination NRT); Test type: Superiority or Other; p = .017, Regression, Logistic; Odds Ratio (OR) = 1.36, 95% CI 2-sided [1.06 to 1.75]
Statistical Analysis 3: Comparison: Standard Cessation Counseling (No CMAC) vs Standard Cessation Counseling Plus CMAC); Null hypothesis: No difference in abstinence rates for participants receiving Standard Cessation Counseling (No CMAC) versus Standard Cessation Counseling plus CMAC. We hypothesized that Standard Counseling plus CMAC would result in statistically significantly higher abstinence rates compared to Standard Counseling Only. The study was originally powered to detect at least a 6.4% increase in the abstinence rate due to an enhanced intervention (e.g., Standard Counseling plus CMAC); Test type: Superiority or Other; p = .343, Regression, Logistic; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.69 to 1.14]

2. Primary Outcome: 7-Day Point Prevalence Abstinence From Smoking by Nicotine Replacement Therapy (NRT) Group
Description: as for outcome 1
Time Frame: 26 weeks after the target quit smoking date
Population: as for outcome 1
Measure: Number; unit: Percentage of participants not smoking
Groups:
- Two Weeks of Nicotine Patch Only: Participants in this treatment group received Two Weeks of Nicotine Patch Only.
- Two Weeks of Combination NRT (Nicotine Patch + Nicotine Gum): Participants in this treatment group received Two Weeks of Nicotine Patch plus Nicotine Gum.
- Six Weeks of Nicotine Patch Only: Participants in this treatment group received Six Weeks of Nicotine Patch Only.
- Six Weeks of Combination NRT (Nicotine Patch + Nicotine Gum): Participants in this treatment group received Six Weeks of Nicotine Patch plus Nicotine Gum.
Arm/Group | Two Weeks of Nicotine Patch Only | Two Weeks of Combination NRT (Nicotine Patch + Nicotine Gum) | Six Weeks of Nicotine Patch Only | Six Weeks of Combination NRT (Nicotine Patch + Nicotine Gum)
Number analyzed (Participants) | 245 | 245 | 249 | 248
Percentage of participants not smoking | 38.4 | 48.2 | 46.2 | 51.6
Statistical Analysis 1: Comparison: Two Weeks of Nicotine Patch Only vs Two Weeks of Combination NRT (Nicotine Patch + Nicotine Gum); Null hypothesis: No difference in abstinence rates for participants receiving Two Weeks of Nicotine Replacement Therapy (NRT) Monotherapy (Nicotine Patch Only) versus Two Weeks of Combination NRT (Patch+Gum). We hypothesized that Two Weeks of Combination NRT would result in statistically significantly higher abstinence rates compared to Two Weeks of NRT Monotherapy. The study was originally powered to detect at least a 6.4% increase in the abstinence rate due to an enhanced intervention; Test type: Superiority or Other; p = .029, Regression, Logistic; Odds Ratio (OR) = 1.49, 95% CI 2-sided [1.04 to 2.14] — Inclusion of the Cognitive Medication Adherence Counseling (CMAC) factor (No CMAC versus CMAC) as a control variable did not change the results of this analysis
Statistical Analysis 2: Comparison: Two Weeks of Nicotine Patch Only vs Six Weeks of Nicotine Patch Only; Null hypothesis: No difference in abstinence rates for participants receiving Two Weeks of Nicotine Replacement Therapy (NRT) Monotherapy (Nicotine Patch Only) versus SIx Weeks of NRT Monotherapy. We hypothesized that Six Weeks of NRT Monotherapy would result in statistically significantly higher abstinence rates compared to Two Weeks of NRT Monotherapy. The study was originally powered to detect at least a 6.4% increase in the abstinence rate due to an enhanced intervention; Test type: Superiority or Other; p = .079, Regression, Logistic; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.96 to 1.97] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Two Weeks of Nicotine Patch Only vs Six Weeks of Combination NRT (Nicotine Patch + Nicotine Gum); Null hypothesis: No difference in abstinence rates for participants receiving Two Weeks of Nicotine Replacement Therapy (NRT) Monotherapy (Nicotine Patch Only) versus Six Weeks of Combination NRT (Patch+Gum). We hypothesized that Six Weeks of Combination NRT would result in statistically significantly higher abstinence rates compared to Two Weeks of NRT Monotherapy. The study was originally powered to detect at least a 6.4% increase in the abstinence rate due to an enhanced intervention; Test type: Superiority or Other; p = .003, Regression, Logistic; Odds Ratio (OR) = 1.71, 95% CI 2-sided [1.20 to 2.45] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Incremental Cost-Effectiveness Ratio for 7-Day Point Prevalence Abstinence From Smoking at 26 Weeks Post-Quit by Nicotine Replacement Therapy (NRT) Group
Description: For cost analyses, we computed the costs of intervention per caller, the cost per quit based on the 6-month ITT 7-day PPA, and the incremental cost-effectiveness ratio (ICER. Intervention costs included direct costs associated with registration, provision of NRT and counseling (standard and MAC), and mailing of a quit guide (all participants) and a MAC information sheet (MAC participants only). Facility space, supplies, and physician supervision time were included in the call costs; research-related costs were excluded. ICER ratio is a measure of the added cost per added quit for two treatments. ICER was computed as the cost difference between the least intensive treatment group (2 weeks of nicotine patch only) and a more intensive comparison group divided by the difference in the quit rates of the two groups being compared; e.g., the ICER for the group that received 2 weeks of nicotine patch and nicotine gum = (213-178)/(.482-.384) = $357.
Time Frame: 26 weeks after the target quit smoking date
Population: No "a priori" power analysis was conducted for this secondary outcome.
Measure: Number; unit: U.S. Dollars
Arm/Group | Two Weeks of Nicotine Patch Only | Two Weeks of Combination NRT (Nicotine Patch + Nicotine Gum) | Six Weeks of Nicotine Patch Only | Six Weeks of Combination NRT (Nicotine Patch + Nicotine Gum)
Number analyzed (Participants) | 245 | 245 | 249 | 248
U.S. Dollars | 94 | 118 | 115 | 128
Statistical Analysis 1: Comparison: Two Weeks of Nicotine Patch Only vs Two Weeks of Combination NRT (Nicotine Patch + Nicotine Gum); In this analysis, the incremental cost-effectiveness ratio (ICER) is computed. ICER is a measure of the added cost per added quit for two treatments. ICER was computed as the cost difference between the least intensive treatment group (2 weeks of nicotine patch only) and a more intensive comparison group divided by the difference in the quit rates of the two groups being compared; ICER for the group that received 2 weeks of nicotine patch and nicotine gum = (213-178)/(.482-.384) = $357; Test type: Superiority or Other; Incremental cost-effectiveness ratio — There is no p-value for the incremental cost-effectiveness ratio (ICER); Unit of measurement for ICER is U.S. dollars; incremental cost-effectiveness ratio = 357
Statistical Analysis 2: Comparison: Two Weeks of Nicotine Patch Only vs Six Weeks of Nicotine Patch Only; In this analysis, the incremental cost-effectiveness ratio (ICER) is computed. ICER is a measure of the added cost per added quit for two treatments. ICER was computed as the cost difference between the least intensive treatment group (2 weeks of nicotine patch only) and a more intensive comparison group divided by the difference in the quit rates of the two groups being compared; ICER for the group that received 6 weeks of nicotine patch only = (233-178)/(.462-.384) = $712; Test type: Superiority or Other; Incremental cost-effectiveness ratio — There is no p-value for the incremental cost-effectiveness ratio (ICER); Unit of measurement for ICER is U.S. dollars; Incremental cost-effectiveness ratio = 712
Statistical Analysis 3: Comparison: Two Weeks of Nicotine Patch Only vs Six Weeks of Combination NRT (Nicotine Patch + Nicotine Gum); In this analysis, the Incremental cost-effectiveness ratio (ICER) is computed. ICER is a measure of the added cost per added quit for two treatments. ICER was computed as the cost difference between the least intensive treatment group (2 weeks of nicotine patch only) and a more intensive comparison group divided by the difference in the quit rates of the two groups being compared; ICER for the group that received 6 weeks of nicotine patch and nicotine gum = (348-178)/(.516-.384) = $1290; Test type: Superiority or Other; Incremental cost-effectiveness ratio — There is no p-value for the incremental cost-effectiveness ratio (ICER); Unit of measurement for ICER is U.S. dollars; Incremental cost-effectiveness ratio = 1290

ADVERSE EVENTS:
Time Frame: Information about adverse events was collected during the 6-week post-quit period of study interventions. The quitline vendor for the study, Free & Clear (Seattle, WA), dispensed all study medications and addressed adverse events.
Description: This study used FDA-approved, over-the-counter nicotine replacement therapies (NRTs) that were dispensed according to standard protocols that were in use by Free & Clear at the time of the study. Free & Clear was responsible for assessing and managing any AEs related to study medication as per their existing Nicotine Replacement Therapy Protocols.
Arm/Group | Two Weeks of Nicotine Patch Only | Two Weeks of Combination NRT (Nicotine Patch + Nicotine Gum) | Six Weeks of Nicotine Patch Only | Six Weeks of Combination NRT (Nicotine Patch + Nicotine Gum)
Serious Adverse Events (participants affected / at risk) | 0/245 | 0/245 | 0/249 | 0/248
Other Adverse Events (participants affected / at risk) | 0/245 | 0/245 | 0/249 | 0/248

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No